CLINICAL TRIAL: NCT00537914
Title: Long-term Phase IV Multicentre Study on the Safety and Efficacy of Omnitrope® (rhGH) in Short Children Born Small for Gestational Age (SGA)
Brief Title: Safety and Efficacy of Omnitrope® (rhGH) in Short Children Born Small for Gestational Age (SGA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP00-401; 2006-002506-58 (EudraCT Number)
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Small for Gestational Age
Keywords: Small for Gestational Age, Omnitrope®/Somatropin, rhGH,SGA
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omnitrope (Experimental): All enrolled patients received Omnitrope. The median daily dose varied between 0.0340 and 0.0351 mg/kg/day and the maximum range was 0.000 to 0.040 mg/kg/day over all visits.
  Interventions: Drug: Omnitrope

INTERVENTIONS:
Drug: Omnitrope — All enrolled patients received Omnitrope. The median daily dose varied between 0.0340 and 0.0351 mg/kg/day and the maximum range was 0.000 to 0.040 mg/kg/day over all visits.
  Other Names: Somatropin

SUMMARY:
This study is performed to investigate the long-term safety, in particular the diabetogenic potential and immunogenicity of rhGH therapy in short children born small for gestational age (SGA).

DETAILED DESCRIPTION:
Prospective, open label, non-comparative, multicenter study. Short children born SGA were to be treated until they reached final height, but treatment could be discontinued earlier if medically indicated or if there was inadequate response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pubertal (Tanner stage I) children born SGA Boys: 4 years of age or older Girls: 4 years of age or older
* Growth disturbance defined as current height SDS < -2.5 (and parental adjusted SDS <-1) for chronological age and sex according to country specific references.
* Birth weight and/or length below -2 standard deviations (SD) for gestational age

Exclusion Criteria:

* Onset of puberty
* Closed epiphyses
* Diabetes mellitus type I or type II
* Fasting blood glucose greater than 100 mg/dl or greater than 5.6 mmol/l measured in venous blood sample
* Abnormal findings in Oral Glucose Tolerance Test (OGTT) defined by greater than 140 mg/dl or greater than 7.8 mmol/l after 120 minutes
* Known IGF-I level above +2SD for sex and age
* Acute critical illness
* Previous treatment with any hGH preparation
* Treatment with antidiabetic medication (e.g. metformin, insulin)
* Drug abuse, substance abuse, or alcohol abuse

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2008-02-06 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz Biopharmaceuticals, Study Chair — Sandoz GmbH
Locations (29):
- Sandoz Investigational Site, Edegem, Antwerpen, Belgium
- Czechia (3):
  - Sandoz Investigational Site, Prague, Prague
  - Sandoz Investigational Site, Hradec Králové
  - Sandoz Investigational Site, Ústí nad Labem
- Sandoz Investigational Site, Tbilisi, Georgia
- Germany (2):
  - Sandoz Investigational Site, Munich, Bavaria
  - Sandoz Investigational Site, Sankt Augustin, North Rhine-Westphalia
- Hungary (4):
  - Sandoz Investigational Site, Szeged, Csongrád megye
  - Sandoz Investigational Site, Budapest
  - Sandoz Investigational Site, Győr
  - Sandoz Investigational Site, Miskolc
- Poland (14):
  - Sandoz Investigational Site, Poznan, Greater Poland Voivodeship
  - Sandoz Investigational Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Sandoz Investigational Site, Wroclaw, Lower Silesian Voivodeship
  - Sandoz Investigational Site, Rzeszów, Podkarpackie Voivodeship
  - Sandoz Investigational Site, Katowice, Silesian Voivodeship
  - Sandoz Investigational Site, Zabrze, Silesian Voivodeship
  - Sandoz Investigational Site, Gdansk
  - Sandoz Investigational Site, Katowice
  - Sandoz Investigational Site, Krakow
  - Sandoz Investigational Site, Lodz
  - Sandoz Investigational Site, Szczecin
  - Sandoz Investigational Site, Warsaw
  - Sandoz Investigational Site, Wroclaw
  - Sandoz Investigational Site, Kielce, Świętokrzyskie Voivodeship
- Romania (4):
  - Sandoz Investigational Site, Cluj-Napoca, Cluj
  - Sandoz Investigational Site, Bucharest
  - Sandoz Investigational Site, Craiova
  - Sandoz Investigational Site, Iași

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was carried out in 31 centers in 7 countries (Poland, Romania, Hungary, Czech Republic, Germany, Belgium and Georgia).
Pre-assignment Details: This study was not randomized. All enrolled patients received Omnitrope
Period: Overall Study
Arm/Group | Omnitrope
Started | 278
Full Analysis Set (FAS) (The FAS followed the ITT principle and comprised all patients who received at least 1 dose of study medication) | 278
Safety Analysis Set (SAS) (The SAF comprised all patients who received at least 1 dose of study medication and had at least 1 post-baseline safety assessment) | 277
Completed | 166
Not Completed | 112
Not completed — Death | 1
Not completed — Adverse Event | 7
Not completed — Treatment failure | 10
Not completed — patients documented other as reason for study discontinuation | 16
Not completed — Lost to Follow-up | 19
Not completed — Withdrawal of informed consent | 59

BASELINE CHARACTERISTICS:
Arm/Group | Omnitrope
Number analyzed (Participants) | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.36 (2.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130
  Male | 148
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 276
  Oriental | 1
  Other: specified as Mixed ethnic origin (Arabic/ Caucasian) | 1
  Black | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Development of Diabetes in Short Children Born SGA During Treatment
Description: The development of diabetes in short children born SGA during treatment was evaluated based on the carbohydrate metabolism parameters FPG, HbA1c and OGTT (basal and 2-h plasma glucose). Only cases which were confirmed by the investigator were included.
Time Frame: throughout the study, approximately 13 years
Population: Safety analysis set: SAF comprised all patients who received at least 1 dose of study medication and had at least 1 post-baseline safety assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Omnitrope
Number analyzed (Participants) | 277
Participants | 0

2. Secondary Outcome: Mean Change in Height (H) (cm) From Baseline
Description: Mean change in Height from baseline for all patients was reported.
Time Frame: Baseline, 3 months, 1 year, 2 years, 5 years and 9 years
Population: Full analysis set: FAS followed the ITT principle and comprised all patients who received at least 1 dose of study medication. Not all patients may have outcome data for all visits.
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Omnitrope
Number analyzed (Participants) | 278
cm
  3 months: number analyzed (Participants) | 276
  3 months | 2.74 [2.62 to 2.86]
  1 year: number analyzed (Participants) | 269
  1 year | 9.08 [8.89 to 9.27]
  2 years: number analyzed (Participants) | 251
  2 years | 16.52 [16.22 to 16.82]
  5 years: number analyzed (Participants) | 211
  5 years | 35.10 [34.48 to 35.72]
  9 years: number analyzed (Participants) | 78
  9 years | 58.07 [56.83 to 59.30]

3. Secondary Outcome: Mean Change in Height Standard Deviation Score Over Time From Baseline
Description: SDS reflects the deviation of a measured value from the mean value of normally growing children of the same sex and chronological age, expressed in units of the standard deviation (SD) of normally growing children of the same sex and chronological age. SDS was calculated according to the formula SDS=(X1-X2)/SD, where X1 is the measured value, X2 the mean value for the relevant chronological age and sex, and SD the reference standard deviation for the relevant sex and age. Refer to SAP page 14 for the formula and to Appendix B (H SDS) and D (HV SDS) for the applied reference Table.
  In general, a negative SDS indicates that the value is below average or mean and a positive value means it is above the average or mean. The calculated mean change compared to baseline reflects the catch-up growth over time towards average normal growth starting from below average.
Time Frame: Baseline, 3 months, 0.5 year, 9 months, 1 year, 1.25 years, 1.5 years, 1.75 years, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years, 11 years, 12 years, 12.5 years
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: SDS
Arm/Group | Omnitrope
Number analyzed (Participants) | 278
SDS
  3 months: number analyzed (Participants) | 276
  3 months | 0.30 [0.28 to 0.33]
  0.5 year: number analyzed (Participants) | 273
  0.5 year | 0.51 [0.47 to 0.54]
  9 months: number analyzed (Participants) | 270
  9 months | 0.68 [0.64 to 0.72]
  1 year: number analyzed (Participants) | 269
  1 year | 0.81 [0.76 to 0.86]
  1.25 years: number analyzed (Participants) | 262
  1.25 years | 0.93 [0.87 to 0.98]
  1.5 years: number analyzed (Participants) | 257
  1.5 years | 1.04 [0.98 to 1.10]
  1.75 years: number analyzed (Participants) | 252
  1.75 years | 1.16 [1.09 to 1.22]
  2 years: number analyzed (Participants) | 251
  2 years | 1.25 [1.18 to 1.31]
  3 years: number analyzed (Participants) | 241
  3 years | 1.50 [1.42 to 1.58]
  4 years: number analyzed (Participants) | 232
  4 years | 1.67 [1.57 to 1.77]
  5 years: number analyzed (Participants) | 211
  5 years | 1.82 [1.70 to 1.94]
  6 years: number analyzed (Participants) | 181
  6 years | 1.94 [1.81 to 2.07]
  7 years: number analyzed (Participants) | 150
  7 years | 2.07 [1.92 to 2.22]
  8 years: number analyzed (Participants) | 118
  8 years | 2.19 [2.03 to 2.35]
  9 years: number analyzed (Participants) | 78
  9 years | 2.18 [1.99 to 2.37]
  10 years: number analyzed (Participants) | 51
  10 years | 2.21 [2.00 to 2.43]
  11 years: number analyzed (Participants) | 28
  11 years | 2.38 [2.13 to 2.63]
  12 years: number analyzed (Participants) | 8
  12 years | 2.39 [1.81 to 2.97]
  12.5 years: number analyzed (Participants) | 3
  12.5 years | 3.01 [1.78 to 4.24]

4. Secondary Outcome: Mean Change in Height Velocity (HV) (cm/Year) Over Time From Baseline
Description: Mean change in Height velocity (HV) (cm/year) over time from baseline was reported.
Time Frame: Baseline, 3 months, 1 year, 2 years, 5 years and 9 years
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: cm/year
Arm/Group | Omnitrope
Number analyzed (Participants) | 278
cm/year
  3 months: number analyzed (Participants) | 276
  3 months | 6.45 [5.95 to 6.95]
  1 year: number analyzed (Participants) | 269
  1 year | 4.71 [4.47 to 4.96]
  2 years: number analyzed (Participants) | 251
  2 years | 3.02 [2.80 to 3.25]
  5 years: number analyzed (Participants) | 211
  5 years | 1.37 [1.01 to 1.73]
  9 years: number analyzed (Participants) | 78
  9 years | 0.10 [-0.53 to 0.74]

5. Secondary Outcome: Mean Change in Height Velocity Standard Deviation Score (HV SDS) Over Time From Baseline
Description: SDS reflects the deviation of a measured value from the mean value of normally growing children of the same sex and chronological age, expressed in units of the standard deviation (SD) of normally growing children of the same sex and chronological age. SDS was calculated according to the formula SDS=(X1-X2)/SD, where X1 is the measured value, X2 the mean value for the relevant chronological age and sex, and SD the reference standard deviation for the relevant sex and age. Refer to SAP page 14 for the formula and to Appendix B (H SDS) and D (HV SDS) for the applied reference Table.
  In general, a negative SDS indicates that the value is below average or mean and a positive value means it is above the average or mean. The calculated mean change compared to baseline reflects the initial high increase in height velocity which remains positive over years, but is decreasing over time.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: SDS
Arm/Group | Omnitrope
Number analyzed (Participants) | 278
SDS
  3 months: number analyzed (Participants) | 276
  3 months | 8.41 [7.76 to 9.07]
  0.5 year: number analyzed (Participants) | 273
  0.5 year | 7.27 [6.83 to 7.71]
  9 months: number analyzed (Participants) | 270
  9 months | 6.69 [6.31 to 7.06]
  1 year: number analyzed (Participants) | 269
  1 year | 6.26 [5.92 to 6.59]
  1.25 years: number analyzed (Participants) | 262
  1.25 years | 5.29 [4.99 to 5.60]
  1.5 years: number analyzed (Participants) | 257
  1.5 years | 4.85 [4.55 to 5.15]
  1.75 years: number analyzed (Participants) | 252
  1.75 years | 4.59 [4.28 to 4.91]
  2 years: number analyzed (Participants) | 251
  2 years | 4.35 [4.02 to 4.68]
  3 years: number analyzed (Participants) | 241
  3 years | 3.62 [3.23 to 4.00]
  4 years: number analyzed (Participants) | 231
  4 years | 3.08 [2.68 to 3.47]
  5 years: number analyzed (Participants) | 211
  5 years | 2.99 [2.50 to 3.49]
  6 years: number analyzed (Participants) | 181
  6 years | 2.63 [2.14 to 3.13]
  7 years: number analyzed (Participants) | 150
  7 years | 2.43 [1.95 to 2.92]
  8 years: number analyzed (Participants) | 118
  8 years | 1.37 [0.75 to 1.98]
  9 years: number analyzed (Participants) | 78
  9 years | 0.85 [0.14 to 1.55]
  10 years: number analyzed (Participants) | 51
  10 years | 0.62 [-0.24 to 1.47]
  11 years: number analyzed (Participants) | 28
  11 years | 1.60 [0.36 to 2.84]
  12 years: number analyzed (Participants) | 8
  12 years | 1.34 [-0.50 to 3.18]
  12.5 years: number analyzed (Participants) | 3
  12.5 years | 1.98 [1.74 to 2.22]

6. Secondary Outcome: Mean Change in Serum IGF-1 Level (Nmol/L) From Baseline
Description: Mean change in serum IGF-1 level (nmol/L) from baseline was reported.
Time Frame: Baseline, 3 months, 1 year, 2 years, 5 years and 9 years
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Omnitrope
Number analyzed (Participants) | 278
nmol/L
  3 months: number analyzed (Participants) | 261
  3 months | 13.04 [11.56 to 14.52]
  1 year: number analyzed (Participants) | 254
  1 year | 20.58 [18.77 to 22.39]
  2 years: number analyzed (Participants) | 234
  2 years | 30.64 [28.16 to 33.12]
  5 years: number analyzed (Participants) | 195
  5 years | 44.87 [41.33 to 48.40]
  9 years: number analyzed (Participants) | 67
  9 years | 75.72 [69.59 to 81.85]

7. Secondary Outcome: Mean Change in IGFBP-3 Levels (Nmol/L) From Baseline
Description: Mean change in IGFBP-3 levels (nmol/L) from baseline was reported.
Time Frame: Baseline, 3 months, 1 year, 2 years, 5 years and 9 years
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Omnitrope
Number analyzed (Participants) | 278
nmol/L
  3 months: number analyzed (Participants) | 250
  3 months | 24.85 [21.64 to 28.05]
  1 year: number analyzed (Participants) | 245
  1 year | 30.48 [27.04 to 33.92]
  2 years: number analyzed (Participants) | 226
  2 years | 48.48 [44.51 to 52.45]
  5 years: number analyzed (Participants) | 189
  5 years | 92.94 [87.65 to 98.23]
  9 years: number analyzed (Participants) | 66
  9 years | 139.12 [126.12 to 152.12]

8. Secondary Outcome: Number of Participants With the Development of Anti-rhGH Antibodies During Omnitrope Treatment
Description: Number of participants with the development of anti-rhGH antibodies with positive test result were reported.
Time Frame: throughout the study, approximately 13 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Omnitrope
Number analyzed (Participants) | 277
Participants | 23

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment to end of the study i.e. up to 13 years.
Description: Any signs or symptoms were collected from first dose of study treatment to end of the study i.e. up to 13 years.
Arm/Group | Omnitrope
All-Cause Mortality (participants affected / at risk) | 1/277
Serious Adverse Events (participants affected / at risk) | 74/277
Other Adverse Events (participants affected / at risk) | 210/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omnitrope (N=277)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Congenital arterial malformation (Congenital, familial and genetic disorders) | 1
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1
Gilbert's syndrome (Congenital, familial and genetic disorders) | 2
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Precocious puberty (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 3
Malabsorption (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Face oedema (General disorders) | 1
Obstruction (General disorders) | 1
Pyrexia (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 4
Bacterial sepsis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Giardiasis (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 2
Infectious mononucleosis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Orchitis (Infections and infestations) | 2
Otitis media (Infections and infestations) | 4
Otitis media acute (Infections and infestations) | 1
Otitis media chronic (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Abdominal injury (Injury, poisoning and procedural complications) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 3
Internal injury (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 2
Traumatic shock (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2
Cardiac murmur (Investigations) | 2
Intraocular pressure increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pachydermodactyly (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain oedema (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Intellectual disability (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 3
Behaviour disorder (Psychiatric disorders) | 1
Enuresis (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Urethral fistula (Renal and urinary disorders) | 1
Urethral stenosis (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Acquired hydrocele (Reproductive system and breast disorders) | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 1
Testicular torsion (Reproductive system and breast disorders) | 2
Varicocele (Reproductive system and breast disorders) | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 1
Circulatory collapse (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omnitrope (N=277)
Hypothyroidism (Endocrine disorders) | 27
Abdominal pain (Gastrointestinal disorders) | 10
Abdominal pain upper (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 13
Pyrexia (General disorders) | 23
Hypersensitivity (Immune system disorders) | 11
Seasonal allergy (Immune system disorders) | 9
Bronchitis (Infections and infestations) | 58
Ear infection (Infections and infestations) | 14
Gastroenteritis (Infections and infestations) | 11
Influenza (Infections and infestations) | 11
Laryngitis (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 78
Otitis media (Infections and infestations) | 19
Otitis media acute (Infections and infestations) | 9
Pharyngitis (Infections and infestations) | 92
Pneumonia (Infections and infestations) | 17
Respiratory tract infection (Infections and infestations) | 25
Rhinitis (Infections and infestations) | 20
Scarlet fever (Infections and infestations) | 11
Sinusitis (Infections and infestations) | 15
Tonsillitis (Infections and infestations) | 35
Upper respiratory tract infection (Infections and infestations) | 47
Urinary tract infection (Infections and infestations) | 17
Varicella (Infections and infestations) | 37
Viral infection (Infections and infestations) | 18
Insulin-like growth factor increased (Investigations) | 9
Scoliosis (Musculoskeletal and connective tissue disorders) | 12
Headache (Nervous system disorders) | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14
Acne (Skin and subcutaneous tissue disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT00537914/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT00537914/SAP_001.pdf